CLINICAL TRIAL: NCT05513053
Title: Immunogenicity and Safety of Quadrivalent Recombinant Influenza Vaccine (RIV4) in Children and Adolescents Aged 9 to 17 Years and Adults Aged 18 to 49 Years.
Brief Title: Study With Quadrivalent Recombinant Influenza Vaccine (RIV4) in Participants 9 Through 49 Years of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAP00027; U1111-1260-4678 (Registry Identifier: ICTRP); VAP00027 (Other: Sanofi Identifier); 2022-000577-11 (EudraCT Number)
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 9 to 17 years old (Experimental): Participants of 9 to 17 years old who received RIV4 single intramuscular (IM) injection at D01
  Interventions: Biological: Quadrivalent Recombinant influenza vaccine (RIV4) season/2022-2023/NH
- Group 18 to 49 years old (Experimental): Participants of 18 to 49 years old who received RIV4 single intramuscular (IM) injection at D01
  Interventions: Biological: Quadrivalent Recombinant influenza vaccine (RIV4) season/2022-2023/NH

INTERVENTIONS:
Biological: Quadrivalent Recombinant influenza vaccine (RIV4) season/2022-2023/NH — Pharmaceutical form: Solution for injection Route of administration: intramuscular
  Other Names: Supemtek / Flublok Quadrivalent

SUMMARY:
The purpose of this study was to demonstrate the non-inferiority (NI) of the HAI immune response of RIV4 in participants aged 9 to 17 years vs participants aged 18 to 49 years and to describe the immunogenicity and safety profile of RIV4 in all participants.

DETAILED DESCRIPTION:
The participation duration was approximately 6 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 49 years on the day of inclusion
* A female participant was eligible to participate if she was not pregnant or breastfeeding and one of the following conditions applies: 1) was of non-childbearing potential. To be considered of non-childbearing potential, a female should have been pre-menarche, post-menopausal for at least 1 year, or surgically sterile OR 2) was of childbearing potential and agreed to use an effective contraceptive method or abstinence from at least 4 weeks prior to the first study intervention administration until at least 4 weeks after the last study intervention administration
* Assent form or informed consent form had been signed and dated by the participant (based on local regulations), and if applicable informed consent form had been signed and dated by the parent(s) or another legally acceptable representative

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination based on the Investigator's judgment
* Personal or family history of Guillain-Barre Syndrome (GBS)
* Personal history of clinically significant development delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder NOTE: The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 9 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1308 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (35):
- United States (21):
  - Alabama Clinical Therapeutics North Tower Site Number : 8400024, Birmingham, Alabama
  - Birmingham Pediatric Associates Site Number : 8400023, Birmingham, Alabama
  - The Children's Clinic Of Jonesboro PA Site Number : 8400025, Jonesboro, Arkansas
  - California Research Foundation Site Number : 8400003, San Diego, California
  - Meridian Clinical Research- Sioux City Site Number : 8400007, Sioux City, Iowa
  - AMR - Newton Site Number : 8400021, Newton, Kansas
  - Kentucky Pediatics / Adult Research Site Number : 8400010, Bardstown, Kentucky
  - Velocity Clinical Research Site Number : 8400012, New Orleans, Louisiana
  - Velocity Clinical Research Lincoln Site Number : 8400013, Lincoln, Nebraska
  - Meridian Clinical Research Norfolk Site Number : 8400011, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha Site Number : 8400009, Omaha, Nebraska
  - Meridian Clinical Research Site Number : 8400006, Binghamton, New York
  - Velocity Clinical Research Vestal Site Number : 8400016, Vestal, New York
  - Ohio Pediatric Research Site Number : 8400020, Dayton, Ohio
  - Rainbow Pediatrics Site Number : 8400014, Barnwell, South Carolina
  - Coastal Pediatric Research Charleston Site Number : 8400005, Charleston, South Carolina
  - Coastal Carolina Research Center - N Charleston Site Number : 8400022, North Charleston, South Carolina
  - Benchmark Research - Austin Site Number : 8400004, Austin, Texas
  - JBR Clinical Research Site Number : 8400001, Salt Lake City, Utah
  - J. Lewis Research Site Number : 8400017, Salt Lake City, Utah
  - Velocity Clinical Research Portsmouth Site Number : 8400015, Portsmouth, Virginia
- Investigational Site Number : 2030001, Jindřichův Hradec, Czechia
- Poland (8):
  - Investigational Site Number : 6160010, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160007, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160004, PuÅ'awy, Lubusz Voivodeship
  - Investigational Site Number : 6160005, Siemianowice Śląskie, Silesian Voivodeship
  - Investigational Site Number : 6160003, Bydgoszcz
  - Investigational Site Number : 6160006, Tarnów
  - Investigational Site Number : 6160008, Warsaw
  - Investigational Site Number : 6160012, Wroclaw
- Spain (5):
  - Investigational Site Number : 7240006, Centelles, Barcelona [Barcelona]
  - Investigational Site Number : 7240018, Madrid
  - Investigational Site Number : 7240005, Málaga
  - Investigational Site Number : 7240001, Móstoles
  - Investigational Site Number : 7240007, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Folegatti PM, Pepin S, Tabar C, Fries K, Talanova O, See S, Essink B, Bertoch T, Drazan D, Natalini Martinez S, Konieczny M, Kaas-Leach K, De Bruijn I. Comparative assessment of immunogenicity and safety of recombinant influenza vaccine in children, adolescents, and adults: results from a phase 3, immunobridging, open-label, non-randomised study. Lancet Infect Dis. 2025 Oct;25(10):1097-1105. doi: 10.1016/S1473-3099(25)00153-7. Epub 2025 May 21. PMID 40412421
- See also: VAP00027 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25371&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 36 investigational sites in 4 countries between 27 Oct 2022 to 27 Oct 2023.
Pre-assignment Details: A total of 1308 participants were enrolled in this study.
Groups:
- Cohort 1: Participants Aged 9 to 17 Years: Participants received a single intramuscular (IM) injection of RIV4 0.5 milliliter (mL) on Day 1.
- Cohort 2: Participants Aged 18 to 49 Years: Participants received a single IM injection of RIV4 0.5 mL on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Started | 648 | 660
Completed | 629 | 635
Not Completed | 19 | 25
Not completed — Lost to Follow-up | 9 | 11
Not completed — Withdrawal by parent/guardian | 2 | 0
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Protocol Violation | 6 | 3
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on study participants with data in case report form (CRF).
Groups:
- Cohort 1: Participants Aged 9 to 17 Years; Cohort 2: Participants Aged 18 to 49 Years: Participants received a single IM injection of RIV4 0.5 mL on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years | Total
Number analyzed (Participants) | 648 | 660 | 1308
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (2.49) | 34.3 (9.21) | 23.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 312 | 395 | 707
  Male | 336 | 265 | 601
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 1 | 6 | 7
  Black or African American | 157 | 98 | 255
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  White | 467 | 536 | 1003
  Not Reported | 0 | 2 | 2
  Unknown | 1 | 1 | 2
  Multiple | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) Against Influenza Vaccine Antibodies at Day 29
Description: GMTs of anti-influenza antibodies were measured using individual hemagglutination inhibition (HAI) assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages.
Time Frame: Day 29
Population: Analysis was performed on the Per-protocol analysis set (PPAS)-subset of full analysis set (FAS) which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 609 | 606
titer
  A/H1N1 | 1946 [1795 to 2109] | 982 [881 to 1094]
  A/H3N2 | 1975 [1771 to 2202] | 604 [531 to 687]
  B/Victoria | 405 [362 to 452] | 258 [233 to 285]
  B/Yamagata | 1941 [1779 to 2118] | 1593 [1477 to 1717]
Statistical Analysis 1: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for A/H1N1; Test type: Non-Inferiority — Non-inferiority was concluded if the lower limit of the two-sided 95% confidence interval (CI) of the ratio of GMTs between groups (9 to 17 years/18 to 49 years) was > 0.667 for each strain; GMT Ratio = 1.98, 95% CI 2-sided [1.73 to 2.27]
Statistical Analysis 2: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for A/H3N2; Test type: Non-Inferiority — Non-inferiority was concluded if the lower limit of the two-sided 95% CI of the ratio of GMTs between groups (9 to 17 years/18 to 49 years) was > 0.667 for each strain; GMT Ratio = 3.27, 95% CI 2-sided [2.76 to 3.87]
Statistical Analysis 3: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for B/Victoria; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.57, 95% CI 2-sided [1.35 to 1.82]
Statistical Analysis 4: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for B/Yamagata; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.22, 95% CI 2-sided [1.09 to 1.37]

2. Primary Outcome: Percentage of Participants With Seroconversion for Influenza Vaccine Antibodies at Day 29
Description: Anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. Seroconversion was defined as either a pre-vaccination titer less than (<) 1:10 (1/dilution) at Day 1 and a post-vaccination titer greater than or equal to (>=) 1: 40 (1/dilution) at Day 29 or a pre-vaccination titer >= 1:10 at Day 1 and a >= 4-fold increase in post-vaccination titer.
Time Frame: Day 29
Population: Analysis was performed on the PPAS-subset of FAS which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category at Day 29 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 609 | 606
percentage of participants
  A/H1N1 | 78.3 [74.8 to 81.5] | 76.4 [72.8 to 79.7]
  A/H3N2 | 86.5 [83.6 to 89.1] | 87.1 [84.2 to 89.7]
  B/Victoria: number analyzed (Participants) | 609 | 605
  B/Victoria | 76.8 [73.3 to 80.1] | 73.6 [69.8 to 77.0]
  B/Yamagata | 77.2 [73.6 to 80.5] | 62.9 [58.9 to 66.7]
Statistical Analysis 1: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for A/H1N1; Test type: Non-Inferiority — Non-inferiority for seroconversion rates was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for the 4 strains; Percent Difference = 1.92, 95% CI 2-sided [-2.78 to 6.62]
Statistical Analysis 2: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for A/H3N2; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percent Difference = -0.59, 95% CI 2-sided [-4.41 to 3.23]
Statistical Analysis 3: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for B/Victoria; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percent Difference = 3.29, 95% CI 2-sided [-1.57 to 8.14]
Statistical Analysis 4: Comparison: Cohort 1: Participants Aged 9 to 17 Years vs Cohort 2: Participants Aged 18 to 49 Years; Statistical analysis for B/Yamagata; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percent Difference = 14.3, 95% CI 2-sided [9.17 to 19.3]

3. Secondary Outcome: GMTs Against Influenza Vaccine Antibodies at Day 1
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages.
Time Frame: Pre-vaccination on Day 1
Population: Analysis was performed on the PPAS-subset of FAS which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category at Day 1 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 609 | 606
titer
  A/H1N1 | 154 [137 to 173] | 74.9 [65.8 to 85.1]
  A/H3N2 | 111 [95.4 to 128] | 29.0 [25.7 to 32.8]
  B/Victoria: number analyzed (Participants) | 609 | 605
  B/Victoria | 48.1 [43.0 to 53.8] | 37.3 [34.0 to 40.9]
  B/Yamagata | 272 [243 to 305] | 300 [269 to 335]

4. Secondary Outcome: Percentage of Participants With Detectable HAI Titers >=10 and >=40 for Influenza Vaccine Antibodies at Days 1 and 29
Description: Antibody titers were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. Percentage of participants with antibody titers >=10 and >=40 against influenza vaccine antibodies at Day 1 and Day 29 were reported in this outcome measure.
Time Frame: On Days 1 and 29
Population: Analysis was performed on the PPAS-subset of FAS which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category on Days 1 and 29 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 609 | 606
percentage of participants
  Titer >=10: A/H1N1: Day 1 | 97.0 [95.4 to 98.2] | 89.8 [87.1 to 92.1]
  Titer >=10: A/H1N1: Day 29 | 100 [99.4 to 100] | 99.3 [98.3 to 99.8]
  Titer >=40: A/H1N1: Day 1 | 87.2 [84.3 to 89.7] | 71.8 [68.0 to 75.3]
  Titer >=40: A/H1N1: Day 29 | 99.7 [98.8 to 100] | 97.5 [96.0 to 98.6]
  Titer >=10: A/H3N2: Day 1 | 89.2 [86.4 to 91.5] | 77.7 [74.2 to 81.0]
  Titer >=10: A/H3N2: Day 29 | 100 [99.4 to 100] | 99.7 [98.8 to 100]
  Titer >=40: A/H3N2: Day 1 | 74.7 [71.1 to 78.1] | 45.0 [41.0 to 49.1]
  Titer >=40: A/H3N2: Day 29 | 99.0 [97.9 to 99.6] | 95.0 [93.0 to 96.6]
  Titer >=10: B/Victoria: Day 1: number analyzed (Participants) | 609 | 605
  Titer >=10: B/Victoria: Day 1 | 92.1 [89.7 to 94.1] | 91.7 [89.2 to 93.8]
  Titer >=10: B/Victoria: Day 29 | 99.5 [98.6 to 99.9] | 99.8 [99.1 to 100]
  Titer >=40: B/Victoria: Day 1: number analyzed (Participants) | 609 | 605
  Titer >=40: B/Victoria: Day 1 | 61.4 [57.4 to 65.3] | 59.8 [55.8 to 63.8]
  Titer >=40: B/Victoria: Day 29 | 95.6 [93.6 to 97.1] | 97.0 [95.3 to 98.2]
  Titer >=10: B/Yamagata: Day 1 | 97.9 [96.4 to 98.9] | 99.5 [98.6 to 99.9]
  Titer >=10: B/Yamagata: Day 29 | 100 [99.4 to 100] | 100 [99.4 to 100]
  Titer >=40: B/Yamagata: Day 1 | 93.1 [90.8 to 95.0] | 95.2 [93.2 to 96.8]
  Titer >=40: B/Yamagata: Day 29 | 99.5 [98.6 to 99.9] | 100 [99.4 to 100]

5. Secondary Outcome: Geometric Mean Titer Ratio (GMTR) of Influenza Vaccine Antibodies
Description: GMTR was the ratio of the individual titers post-vaccination over pre-vaccination. The GMTs were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages.
Time Frame: On Days 1 and 29
Population: Analysis was performed on the PPAS-subset of FAS which included participants who received 1 dose of the study vaccine and had a post-vaccination blood sample. Only participants with data collected for each category on Days 1 and Day 29 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 609 | 606
ratio
  A/H1N1 | 12.7 [11.1 to 14.5] | 13.1 [11.4 to 15.0]
  A/H3N2 | 17.9 [15.7 to 20.3] | 20.8 [18.4 to 23.6]
  B/Victoria: number analyzed (Participants) | 609 | 605
  B/Victoria | 8.41 [7.55 to 9.37] | 6.91 [6.25 to 7.64]
  B/Yamagata | 7.13 [6.46 to 7.87] | 5.31 [4.79 to 5.88]

6. Secondary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, that is, prelisted in the CRF in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs.
Time Frame: Within 30 minutes post-vaccination on Day 1
Population: Analysis was performed on the Safety analysis set which included participants who received 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 641 | 658
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted in the protocol and CRF and considered as related to the study intervention administered. An injection site reaction was an AR at and around the injection site and were commonly inflammatory reactions. Solicited systemic reactions were systemic AEs and those occurring during the specified collection period were always considered related to the intervention even if there was evidence of alternative etiology.
Time Frame: From Day 1 up to 7 days post-vaccination (up to Day 8)
Population: Analysis was performed on the Safety analysis set which included participants who received 1 dose of the study vaccine. Number of participants analyzed signifies those participants with data collected for this outcome measure and number analyzed signifies those participants with data collected for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 618 | 635
Participants
  Solicited injection site reaction | 220 | 259
  Solicited systemic reaction: number analyzed (Participants) | 615 | 635
  Solicited systemic reaction | 182 | 230

8. Secondary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, that is, prelisted in the CRF in terms of diagnosis and/or onset window post-vaccination.
Time Frame: From Day 1 up to 28 days post-vaccination (up to Day 29)
Population: Analysis was performed on the Safety analysis set which included participants who received 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 641 | 658
Participants | 93 | 119

9. Secondary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs)
Description: An MAAE was a new onset or a worsening of a condition that prompted the participant or participant's parent/guardian to seek unplanned medical advice at a physician's office or emergency department.
Time Frame: From Day 1 up to 28 days post-vaccination (up to Day 29)
Population: Analysis was performed on the Safety analysis set which included participants who received 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 641 | 658
Participants | 27 | 35

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) And Adverse Events of Special Interest (AESI)
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI was defined as one of scientific and medical concern specific to the Sponsor's study intervention, events for which ongoing monitoring and rapid communication by the investigator to the sponsor was done.
Time Frame: From Day 1 up to 6 months post-vaccination, 181 days
Population: Analysis was performed on the Safety analysis set which included participants who received 1 dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
Number analyzed (Participants) | 641 | 658
Participants
  SAE | 3 | 7
  AESI | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to 6 months post-vaccination, 181 days
Description: Analysis was performed on the Safety analysis set.
Arm/Group | Cohort 1: Participants Aged 9 to 17 Years | Cohort 2: Participants Aged 18 to 49 Years
All-Cause Mortality (participants affected / at risk) | 0/641 | 0/658
Serious Adverse Events (participants affected / at risk) | 3/641 | 7/658
Other Adverse Events (participants affected / at risk) | 263/641 | 336/658
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Participants Aged 9 to 17 Years (N=641) | Cohort 2: Participants Aged 18 to 49 Years (N=658)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastric Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 2 (3) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Participants Aged 9 to 17 Years (N=641) | Cohort 2: Participants Aged 18 to 49 Years (N=658)
Headache (Nervous system disorders) | 114 (121) | 152 (153)
Myalgia (Musculoskeletal and connective tissue disorders) | 119 (119) | 129 (129)
Chills (General disorders) | 45 (45) | 40 (40)
Injection Site Pain (General disorders) | 212 (212) | 255 (256)
Malaise (General disorders) | 100 (100) | 106 (106)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT05513053/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT05513053/SAP_001.pdf